CLINICAL TRIAL: NCT04338932
Title: COVID-19 and Deep Venous Thrombosis: a Cross-sectional Study
Brief Title: COVID-19 and Deep Venous Thrombosis
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Dr, Jessa Hospital
Other Study IDs: JessaH_COVID19_DVT
Record Dates: First submitted 2020-04-07; First posted 2020-04-08 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Deep Vein Thrombosis (DVT)/Thrombophlebitis
MeSH Terms: conditions — COVID-19; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the prevalence and possible risk factors of the occurrence of a DVT in 12 intubated and mechanically ventilated COVID-19 patients admitted to the ICU at a single time point (29/03/2020).

DETAILED DESCRIPTION:
Patients admitted to the Intensive Care Unit (ICU) are known to be at risk for thrombo-embolic events. Virchow's triad describes the major risk factors in three categories: venous stasis, vessel injury and activation of blood coagulation. A prolonged mechanical ventilation together with the hemodynamic effects of this ventilation with a high positive and expiratory pressure (PEEP), the presence of central venous catheters, the immobilization of these patients and the presence of obesity or other comorbidities can attribute to the occurrence of a deep venous thrombosis (DVT) in patients admitted at ICU. The incidence of DVT during ICU stay has been reported between 5 and 15%.

On the 13th of March, the first COVID-19 patient was admitted at the ICU at the Jessa Hospital. Within a few days, the admissions at our COVID-19 unit grew exponential. In these difficult time, research concerning COVID-19 has been performed indicating the COVID-19 virus induces a hyper-inflammatory state. It has been suggested that systemic inflammation induces endothelial injury. This will activate the coagulation cascade and impair fibrinolysis with disruption of endothelial barrier, and loss of physiologic antithrombotic factors which may elevated the risk for DVTs significantly. Up to now, there is still no causal treatment for COVID-19. The current management of COVID-19 is mainly supportive i.e. a prolonged inflammatory status and a prolonged risk for VTE.

During the placement of a dialysis catheter in the femoral vein of one of the patients admitted in the ICU for COVID-19 at our hospital, a large deep vein thrombosis (DVT) proximal in both common femoral veins was noticed in a patient. Since there were no clinical signs of DVT present in this patient, every patient at the ICU unit at that moment was screened on the presence of DVTs. We found one or several deep vein thromboses in 8 out of 12 patients at 1 ICU unit. Since this was a unusual high incidence, we want to further investigate this prevalence and evaluate possible causes of these DVTs.

The aim of this study is to investigate the prevalence and possible risk factors of the occurrence of a DVT in 12 intubated and mechanically ventilated COVID-19 patients admitted to the ICU at a single time point (29/03/2020).

The endpoint of this cross-sectional study is to investigate the prevalence and identify possible risk factors of the occurrence of a DVT in these patients at the ICU.

These parameters are listed below and included parameters/values collected as a standard-of-care in our hospital:

* Demographics: i.e age, gender
* Comorbidities: smoking, hypertension, diabetes, cardiovascular disease, respiratory disease, malignancies, renal failure, liver failure, gastrointestinal disease, neurological conditions, mental state, other
* Symptoms at the time of admission to ICU: i.e fever, body temperature, dyspnoea, headache, diarrhea etc…
* Laboratory results of all standard parameters measured
* Treatment: antiviral agents, antibiotics, etc…
* Complications: shock, heart failure, sepsis, stroke, etc…
* Ventilation: method, PEEP, FiO2, ..
* Radiological findings: pneumonia, ground-glass opacity..

ELIGIBILITY:
Inclusion Criteria:

* 12 intubated and mechanically ventilated COVID-19 patients admitted to the ICU at a single time point (29/03/2020).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 12 intubated and mechanically ventilated COVID-19 patients admitted to the ICU at a single time point (29/03/2020).
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
the prevalence of a DVT in patients at the ICU. | 1 day at ICU
  to investigate the prevalence of a DVT in patients at the ICU.

SECONDARY OUTCOMES:
Oxygen partial pressure and Carbon dioxide partial pressure levels in the blood | 1 day at ICU
  evaluate pO2 and pCO2 (mmHg) in patients with and without a DVT
Potassium, Sodium, Calcium, Bicarbonate, Base excess, Lactate levels in the blood | 1 day at ICU
  evaluate Potassium, Sodium, Calcium, Bicarbonate, Base excess, Lactate levels (mmol/l) in patients with and without a DVT
glucose, haemoglobin, ureum, creatinine, total bilirubin levels in the blood | 1 day at ICU
  evaluate glucose, haemoglobin, ureum, creatinine, total bilirubin levels (mg/dl) in patients with and without a DVT
oxygen saturation, basophils, eosinophils, monocytes, neutrophils, haematocrit and prothrombine levels in the blood | 1 day at ICU
  evaluate oxygen saturation, basophils, eosinophils, monocytes, neutrophils, haematocrit and prothrombine levels in the blood (%) in patients with and without a DVT
white blood cells, red blood cells and platelets in the blood | 1 day at ICU
  evaluate white blood cells (x 10*9/L), red blood cells (x 10*12/L) and platelets levels (x 109/L) in the blood in patients with and without a DVT
PT (%)aPTT (sec)Fibrinogen (g/L)D-dimers (mg/L) PT (INR) (ratio) AST (U/L)ALT (U/L)Lactate dehydrogenase (U/L)Troponin T (ng/L)CRP (mg/L)Ferritin (mg/L)in the blood | 1 day at ICU
  evaluate PT (%)aPTT (sec)Fibrinogen (g/L)D-dimers (mg/L) PT (INR) (ratio) AST (U/L)ALT (U/L)Lactate dehydrogenase (U/L)Troponin T (ng/L)CRP (mg/L)Ferritin (mg/L) in the blood in patients with and without a DVT
prevalence of co-morbidities | 1 day at ICU
  revalence of co morbidities such as Cardiovascular disease, n (%) Hypertension, n (%) Diabetes, n (%) Respiratory disease, n (%) Malignancy, n (%) Chronic renal disease, n (%) Chronic liver disease, n (%) Chronic bowel disease, n (%) Chronic nerve disease, n (%) Cerebrovascular disease, n (%) HIV/AIDS, n (%) Haematological disease, n (%) Obesity, n (%) Rheumatological disease, n (%) Dementia, n (%) in patients with and without a DVT admitted at the ICU in 1 day
prevalence of vital signs at icu admission | at ICU admission
  prevalence of vital signs such Temperature (°C) Breathing rate (#/min) Systolic blood pressure (mmHg) Mean arterial blood pressure (mmHg) Heart rate (#/min) Glasgow Coma Scale in patients with and without a DVT
prevalence of complications during icu stay | from ICU admission to cross sectional moment (29/3/2020)
  prevalance of complications such as ARDS Acute kidney failure Acute heart failure Septic shock Secondary infection Seizure Stroke Hyperglaecemia Hypoglaecemia during ICU stay in patients with and without DVT
evaluation of treatment | from ICU admission to cross sectional moment (29/3/2020)
  evaluation of treatment such as Antiviral treatment Antibiotic treatment Antifungal treatment Corticosteroid treatment CRRT IVIg treatment Plaquenil treatment during ICU stay in patients with and without DVT
evaluation of the oxygen therapy | from ICU admission to cross sectional moment (29/3/2020)
  evaluation of the oxygen therapy such as Invasive mechanical ventilation FiO2 (mmHg) PEEP Length of ventilationA ECMO Invasive mechanical ventilation + ECMO Vasopressor/inotropic support Neuromuscular blocking agents Prone ventilation in patients with and without DVT

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No